CLINICAL TRIAL: NCT03872271
Title: Is Diverting Loop Ileostomy Necessary in Completion Proctectomy With Ileal Pouch Anal- Anastomosis: A Multicentre, Randomized Study of the GETAID Chirurgie Group. IDEAL Trial
Acronym: IDEAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-04; 2019-A00687-50 (Other: IDRCB number)
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Ulcerative Colitis; Ileostomy - Stoma
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Proctocolectomy, Restorative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): ileal pouch-anal anastomosis without diverting loop ileostomy
  Interventions: Procedure: ileal pouch-anal anastomosis with diverting loop ileastomy
- Control (Active Comparator): ileal pouch-anal anastomosis with diverting loop ileostomy
  Interventions: Procedure: ileal pouch-anal anastomosis with diverting loop ileastomy

INTERVENTIONS:
Procedure: ileal pouch-anal anastomosis with diverting loop ileastomy — Defunctioning ileostomy has demonstrated its benefits (rate and seriousness of anastomotic leakage) in cancer for low colorectal and coloanal anastomoses, whereas there are no such good quality evidences in case of ileal pouch-anal anastomosis (IPAA) performed for inflammatory bowel disease (IBD). However, most surgical teams do protect systematically IPAA by an ileostomy.
  Arms: Control
Procedure: ileal pouch-anal anastomosis with diverting loop ileastomy — Defunctioning ileostomy has demonstrated its benefits (rate and seriousness of anastomotic leakage) in cancer for low colorectal and coloanal anastomoses, whereas there are no such good quality evidences in case of ileal pouch-anal anastomosis (IPAA) performed for inflammatory bowel disease (IBD). However, most surgical teams do protect systematically IPAA by an ileostomy.
  Arms: Experimental

SUMMARY:
Defunctioning ileostomy has demonstrated its benefits (rate and seriousness of anastomotic leakage) in cancer for low colorectal and coloanal anastomoses, whereas there are no such good quality evidences in case of ileal pouch-anal anastomosis (IPAA) performed for inflammatory bowel disease (IBD). However, most surgical teams do protect systematically IPAA by an ileostomy.

Total proctocolectomy with IPAA is the gold standard for surgical management of ulcerative colitis (UC). This demanding procedure is often performed in 2 or 3 stages, namely subtotal colectomy, completion proctectomy with IPAA and defunctioning ileostomy closure. Subtotal colectomy with double stoma is first performed to allow nutritional support, reduce inflammation and stop immunosuppressive agents. Completion proctectomy with IPAA is then performed on a healthier patient. Hence, the need for a systematic defunctioning ileostomy is questioned. No study addressed specifically the question of completion proctectomy, whereas it concerns 36% to 42% of patients undergoing IPAA. Globally, the overall 6-month morbidity rate is 55% in case of stoma creation vs. 30% otherwise in IPAA.

Moreover, defunctioning ileostomy has several drawbacks including an additional surgical procedure (stoma closure), a worse quality of life before closure, and the risk of dehydration that may require readmission. Following stoma closure, the risk of anastomotic leakage is around 4%. Overall, during the stoma period, 8% of patients will require reoperation. Finally, the risk of incisional hernia is 15-20% at the ex-ileostomy site.

Therefore, the aim of this trial is to assess the need for a systematic defunctioning ileostomy after completion proctectomy with IPAA.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥ 18 years,
* patients presenting with ulcerative colitis or indeterminate colitis requiring completion proctectomy
* patients who have given informed consent

Exclusion Criteria:

* indication for total proctocolectomy in one-stage or traditional 2-stage fashion
* Crohn's disease,
* pelvic radiotherapy,
* indication for total mésorectum excision
* vulnerable patient under the French laws

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2024-05-24 (Estimated); Study Completion 2025-05-24 (Estimated)

PRIMARY OUTCOMES:
6-month global postoperative morbidity | 6 months
  Number and qualification of surgical and medical complications that may require redmission during the 6 months following the operative procedure:
  * SBO
  * ileostomy prolapse
  * parastomial hernia
  * dehydration
  * skin erosions, that may require readmission
  * anastomotic leakage
  * incisional hernia.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — AP-HM
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beyer-Berjot L, Baumstarck K, Loubiere S, Vicaut E, Berdah SV, Benoist S, Lefevre JH; GETAID Chirurgie group. Is diverting loop ileostomy necessary for completion proctectomy with ileal pouch-anal anastomosis? A multicenter randomized trial of the GETAID Chirurgie group (IDEAL trial): rationale and design (NCT03872271). BMC Surg. 2019 Dec 12;19(1):192. doi: 10.1186/s12893-019-0657-7. PMID 31830976